CLINICAL TRIAL: NCT02158585
Title: Lamotrigine for Ménière's Disease: a Double-blind, Placebo-controlled Pilot Study
Brief Title: Study of Lamotrigine to Treat Ménière's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dent Neuroscience Research Center (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Principal Investigator, Lixin Zhang, Medical Director of the Dizziness and Balance Center, Dent Neuroscience Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Zhang-001
Record Dates: First submitted 2014-06-02; First posted 2014-06-09 (Estimated); Results first posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-05

CONDITIONS: Meniere's Disease; Ménière's Vertigo; Vertigo, Intermittent; Vertigo, Aural
Keywords: Lamotrigine; Lamictal; Anticonvulsant; Ménière's disease; Vertigo attack; Dizziness; Vestibular disorder
MeSH Terms: conditions — Meniere Disease; Vertigo; Dizziness; Vestibular Diseases | interventions — Lamotrigine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo will match the lamotrigine dosage, frequency and duration.
  Interventions: Drug: Placebo
- Lamotrigine (Active Comparator): Lamotrigine will be taken orally for the duration of 20 weeks, consisting of a six-week titration, 12-week study period, and two-week taper. Possible doses are 25mg twice a day, 50mg twice a day, and 100 mg twice a day during titration; 150mg twice a day for the 12-week study period; 150mg once a day for Week 1 of the taper; and 75mg once a day for Week 2 of the taper. Patients who withdraw at any point of the study will have a two-week taper consisting of the current dose once a day for one week followed by half the dose once a day for another week.
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lamotrigine — Lamotrigine will be taken orally on a daily basis for the duration of 20 weeks, consisting of a six-week titration, 12-week study period, and two-week taper. Possible doses for patients are 25mg twice a day, 50mg twice a day, and 100 mg twice a day during titration; 150mg twice a day for the 12-week study period; 150mg once a day for Week 1 of the taper; and 75mg once a day for Week 2 of the taper. Each increase in dose will be maintained for two weeks before deciding to further increase or decrease based on tolerability. Patients who discontinue at any point of the study will have a two-week taper consisting of the current dose once a day for one week followed by half the dose once a day for another week.
  Other Names: Lamictal; 3,5-diamino-6-(2,3-dichlorophenyl)-as-triazine; U3H27498KS
  Arms: Lamotrigine
Drug: Placebo — The placebo will match the lamotrigine dosage, frequency and duration.
  Other Names: microcrystalline cellulose
  Arms: Placebo

SUMMARY:
This double-blinded study evaluates the frequency of vertigo attacks and the quality of life of patients diagnosed with Ménière's disease after being randomly assigned to take a placebo or lamotrigine.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 years or older
* Diagnosed with unilateral definite Ménière's disease according to the AAO-HNS 1995 criteria, confirmed by an ENT
* Active vertigo: at least two Ménière's vertigo attacks (defined as lasting 20 minutes or longer and associated with tinnitus, ear fullness, or low frequency hearing loss and nausea/vomiting) every four weeks during the eight-week qualification period and at least two more Ménière's vertigo attacks during the lead-in phase prior to randomization
* Documented unilateral lower frequency hearing loss defined as the four-tone average (arithmetic mean rounded to the nearest whole number) of the pure-tone thresholds at 0.25, 0.5, 1 and 2 kilohertz (kHz) more than or equal to 25 decibels (dB) of the worse audiogram during the six months before screening
* Have tried diuretics for at least one month and discontinued treatment due to continued vertigo attacks
* All other co-existing medical or psychiatric conditions are stable, and no greater than moderate severity
* Willing to avoid pregnancy during the entirety of the study (abstinence or two forms of acceptable birth control, such as condoms and oral contraceptives)

Exclusion Criteria:

* Bilateral Ménière's disease
* Current or past history of migraine
* Any other neuro-otologic disease or major vestibular abnormality found during screening that could confound the evaluation of Ménière's symptoms
* Previous intolerance or sensitivity to lamotrigine
* On any prohibited medication within four weeks prior to the study
* History of tympanostomy tubes with evidence of perforation or lack of closure
* IT gentamicin injections or endolymphatic sac surgery within the last year
* History of or current immunodeficiency disease, nephrolithiasis, hypertension, cardiac disease, arrhythmia, hypercholesterolemia, hemiplegic/basilar migraine, stroke, diabetes, vascular disease or kidney disease
* Family history of unexplained deafness
* Pregnant or breastfeeding
* Current diseases or conditions that may be associated with an altered perception of processing stimuli
* Current severe medical condition(s) that in the view of the investigator prohibits participation
* Previously used the investigational drug
* Current non-vertiginous dizziness (orthostatic or panic disorder) unless it could be clearly differentiated from Ménière's attacks by the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Zhang, MD, PhD, Principal Investigator — Dent Neurologic Institute
Locations (1):
- Dent Neurologic Institute, Amherst, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12-week pre-treatment period
Period: Overall Study
Arm/Group | Placebo | Lamotrigine
Started | 8 | 7
Completed | 7 | 6
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lamotrigine | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (13.8) | 55.1 (12.9) | 57.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 2 | 4 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Ménière's Vertigo Attack Frequency Between Lamotrigine and Placebo Group
Description: Measured with a daily questionnaire
Time Frame: Duration of 12-week pre-treatment and 12-week study period (treatment)
Measure: Mean (Standard Deviation); unit: Average Total Number of Vertigo Attacks
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 8 | 7
Average Total Number of Vertigo Attacks
  Pre-Treatment (Week -12 to -1) | 18.88 (6.27) | 18.00 (12.65)
  Treatment (Week 7 to 18) | 13.50 (14.54) | 4.57 (4.96)
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine; Null hypothesis: no difference between groups in average total number of vertigo attacks; Test type: Superiority; p = 0.5618, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 8.93, 95% CI 2-sided [-3.49 to 21.35]

2. Primary Outcome: Change in Ménière's Vertigo Attack Frequency Within Lamotrigine Group
Description: Measured with daily questionnaire
Time Frame: Duration of 12-week pre-treatment and 12-week study period (treatment)
Measure: Mean (Standard Deviation); unit: Average Total Number of Vertigo Attacks
Arm/Group | Lamotrigine
Number analyzed (Participants) | 7
Average Total Number of Vertigo Attacks
  Pre-treatment | 18.00 (12.65)
  Study Period | 4.57 (4.96)
Statistical Analysis 1: Comparison: Lamotrigine; Null hypothesis: no difference between average total number of vertigo attacks in pre-treatment and treatment; Test type: Superiority; p = 0.03429, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Difference in Ménière's Vertigo Attacks in Three-Week Intervals Between Lamotrigine and Placebo Groups
Description: Measured with a daily questionnaire.
Time Frame: Duration of Week 16 to 18
Measure: Mean (Standard Deviation); unit: Average Total Number of Vertigo Attacks
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 8 | 7
Average Total Number of Vertigo Attacks | 4.86 (4.02) | 0.29 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine; Null hypothesis: no difference in total average number of vertigo attacks during 3 week time periods; Test type: Superiority; p = 0.0092, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 4.57, 95% CI 2-sided [0.85 to 8.29]

4. Secondary Outcome: Improvement in Pure Tone Average in the Affected Ear
Description: Measured using the average of 500, 1000, 2000, and 3000 Hz presentation level (dB)
Time Frame: Prior to randomization and at completion of 12-week study period
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 8 | 7
Participants | 3 | 5

5. Secondary Outcome: Improvement in Symptoms Severity
Description: Based of rating on Clinical Global Impression of Change (CGI) score of blinded physician
Time Frame: 12-week pre-treatment period; 6 week titration; 12-week study period (treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 8 | 7
Participants | 3 | 6

6. Secondary Outcome: DHI Scores
Description: Dizziness Handicap Inventory (DHI). Minimum score=0. Maximum score=100. Higher scores mean a worse outcome.
Time Frame: Baseline (Week 1) and end of study (Week 18)
Measure: Mean (Standard Deviation); unit: score on DHI
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 8 | 7
score on DHI
  Baseline | 57.50 (17.26) | 37.14 (12.05)
  End of Study | 49.43 (25.73) | 38.29 (19.44)
Statistical Analysis 1: Comparison: Placebo vs Lamotrigine; Test type: Superiority; p = 0.0385, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 11.14, 95% CI 2-sided [-15.64 to 37.92]

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: Patients reported whether or not there were any changes in health during every study visit. They were also encouraged to call the clinic if there were any changes.
Groups:
- Lamotrigine: Lamotrigine will be taken orally for the duration of 20 weeks, consisting of a six-week titration, 12-week study period, and two-week taper. Possible doses are 25mg twice a day, 50mg twice a day, 100 mg twice a day and 150mg twice a day during titration; 150mg twice a day or 100mg twice a day for the 12-week study period; 150mg once a day, or 100mg once a day for Week 1 of the taper; and 75mg once a day, or 50mg once a day for Week 2 of the taper. Patients who withdraw at any point of the study will have a two-week taper consisting of the current dose once a day for one week followed by half the dose once a day for another week.
Arm/Group | Placebo | Lamotrigine
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | Lamotrigine (N=7)
Gastrointestinal problem (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02158585/Prot_SAP_000.pdf